CLINICAL TRIAL: NCT03233828
Title: Pre-Treatment of Highly Suspicious Pigmented Skin Lesions With Interleukin-2
Acronym: IL-2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment numbers.
Sponsor: Carman Giacomantonio (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Carman Giacomantonio, Surgical Oncologist / General Surgeon / Professor, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4387
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Melanoma (Skin); Melanoma in Situ
Keywords: Intralesional Injection; Immunotherapy; Immune Response; Interleukin-2 (Aldesleukin); Tumor Infiltration; Metastasis Prevention
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be given either intralesional IL-2 or intralesional saline as a control
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intralesional IL-2 Injection (Experimental): Two subcutaneous intralesional injections of Aldesleukin, prepared by the pharmacy such that the contents will be masked, will be administered by the care provider in a clinic seven days apart.
  Interventions: Biological: Aldesleukin
- Saline Injection (Placebo Comparator): Two subcutaneous intralesional injections of Saline, prepared by the pharmacy such that the contents will be masked, will be administered by the care provider in a clinic seven days apart.
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Aldesleukin — 500,000 IU in 0.1mL
  Arms: Intralesional IL-2 Injection
Other: Saline — 0.1 mL of sterile saline solution (0.9% m/v)
  Arms: Saline Injection

SUMMARY:
This study is meant to assess the use of intralesional IL-2 to modulate the immunological response to suspected melanoma, or melanoma in situ, in an effort to increase lymphocyte infiltration and decrease disease metastasis.

Patients that are clinically diagnosed with suspected Melanoma or Melanoma in situ will be assigned to either a treatment or control arm. The treatment group will be subjected to two intralesional IL-2 injections, whereas the control group will be subjected to two intralesional injections of saline.

The proteomic and metabolomic profiles of both groups will be analyzed using urine and blood samples in an effort to assess the systemic immunological response, if any, to the treatment. Also, upon disease confirmation and staging by a qualified pathologist, lesions will be assessed for lymphocyte infiltration using immunohistochemical methods.

This study will determine whether pre-treatment of IL-2 on lesions (clinically diagnosed as melanoma or melanoma in situ) is effective in generating an adaptive immune response, and whether that immune response may play a role in preventing disease metastasis.

DETAILED DESCRIPTION:
This study is primarily designed to determine if tumor specific immunity can be generated in patients with highly suspicious pigmented lesions in response to intralesional IL-2, and whether that immunity can confer resistance to melanoma metastasis. Patients will be identified by qualified dermatologists and interviews will be held at the surgery clinic (4th floor Dickson Center) QEII HSC, NSHA.

The standard wait time from consultation to surgical biopsy is up to 4 weeks. Investigators will ensure that patients are seen immediately upon notification from participating dermatologist and all research components of the study are completed within the normally anticipated wait time. Through utilization of this standard wait time, intralesional IL-2 can potentially affect an immune response, that otherwise could not be achieved after the biopsy is completed. Given that the study is conducted within the normal wait time, it doesn't deviate from the normal standard of care. Following the study protocol, patients will receive intralesional injections on Day 1(Week 1 Visit) and Day 8 (Week 2 Visit), and excisional biopsies will be performed on Day 15 (Week 3 Visit), well within the accepted wait time from consultation to biopsy. The intralesional injections and collection of biospecimens beyond the biopsy deviate from but does not delay the normal standard of care. Two additional visits are required in addition to the initial consultation.

This study is a randomized, controlled, double-blind study. Patients with highly suspicious pigmented lesions will be randomly assigned by an algorithm to one of two groups: 1) treatment group patients will be treated intralesionally with IL-2 (Proleukin (Aldesleukin), Novartis Pharmaceuticals Canada Inc.) at a dose of 500,000 International Units (IU) in 0.1ml of sterilized saline (0.9%, m/v) for 2 treatment cycles 1 week apart (Day 1 and Day 7); 2) control group patients will be treated intralesionally with sterilized saline (0.9%, m/v) of the same volume (0.1ml). Randomization will be generated by a Random Block algorithm for each patient, and instruction preparation for each patient will be sent to pharmacy. IL-2 (Proleukin) will be obtained from Novartis by the pharmacy, paid for by Dr. Carman Giacomantonio's research services account. The pharmacy will be given instruction to prepare either IL-2 treatment or injectable control (saline). The pharmacy will assign a codified ID which will be provided along with the syringe with the patient name labeled as "Interleukin-2/Placebo" (thus blinding study to clinician and patient). As a pilot study, the principle of the design is to test the feasibility of proceeding to a larger and more expensive trial following the methodology and protocol proposed. As such there will be a minimum of 20 (10 treatment, 10 placebo) participants (up to a maximum of 60). It is estimated that statistical significance will be reached with 20 patients, however if it is not reached after 20 patients, an additional 10 (5 treatment, 5 control) patients will be enrolled. If significance is still not reached after 30 patients, an additional 10 patients will be enrolled and so on up to a maximum of 60 patients. If after 60 patients, significance is not achieved then further recruitment under the current protocol would not be logical and therefore the methodology would need to be revised or study discontinued.

On Day 1 (first treatment) and 15 (excisional biopsy), all patients will have blood (4 vials) and urine (25-50 ml) samples taken. Local reactions to injections will be monitored for non- specific signs such as bleeding, arythema, infection, or irritation. Investigators do not anticipate specific changes in the pigmented lesion related to the injection in this short time period, however all changes will be noted.

On Day 15, following the second intralesional injection an excisional biopsy will be performed following standard surgical techniques, as follows: ellipse of skin encompassing the pigmented lesion extending into the subcutaneous fat will be performed to achieve a grossly clear but narrow margin of excision. This small defect will be closed primarily with interrupted sutures. The biopsied specimen will be subsequently evaluated using standard histological techniques to confirm diagnoses, assess margin status (clear or involved) and depth of lesion invasion. The depth of lesion invasion will dictate the extent of subsequent surgical excisions and margin selection according to standard National Comprehensive Cancer Network (NCCN) guidelines. Pre-biopsy intralesional injections of 0.1ml into the lesion will not alter dimensions or architecture of the lesion or impact the extent the subsequent biopsy required. Lesions that are felt to be too large for closure without tissue manipulation or creation of flaps, will be biopsied using a punch biopsy sampling technique whereby 4mm diameter discs of tissue from representative areas of the lesion will be taken to confirm the diagnosis and the depth of invasion. The depth of invasion will dictate the extent and complexity of subsequent surgery required to remove the lesion and achieve clear margins according to NCCN guidelines. The biopsied specimen will be processed as follows: using a 22G needle a fine needle aspiration biopsy will be performed (the needle will be passed through the center of the lesion two times) for RNA analysis. The remainder of the tissue will be sent to pathology for standard histological assessment. The pathologist will also report the extent of observed tumor infiltrating lymphocytes (TILs) associated with treatment compared to control injections. Blood and urine will be assessed using metabalomic and proteomic methods to assess systemic immune response to treatment.

All blood, urine, and lesion biopsy samples will be labeled with a codified number (will not contain any patient identifying information) and will be immediately transported to Dr. Carman Giacomantonio laboratory at Dalhousie University for storage. Fine needle aspiration of excised samples will be assessed for tumor genetic and epigeneitic profile. Blood and urine will be assessed for proteomic and metabolomic profiles, respectively.

All study participants will receive assessments every 4 months for 2 years and biannual assessments for years 3 to 5 after the initial intervention to assess disease progression, or the development of new melanoma, to compare between both treatment and control groups. There is no standardize test or measurable biomarker to assess established or lasting immunity. This aspect of the study is identical to the patient assessment conducted as per standard of care for melanoma patients. Again, any publications of study results will be completed devoid of any information that could be used to identify patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

* The participant population will include patients characterized by: nodular/polypoid features, bleeding/ulcerated lesions, excluding face and vulvo-genital lesions.

Exclusion Criteria:

* Participants who are not: currently immunocompromized, on immuno-therapy for other diagnosis, have known inflammatory or autoimmune diseases or are otherwise incapacitated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carman A Giacomantonio, MD, FRCSC, Principal Investigator — Surgical Oncologist / General Surgeon / Professor
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranieri JM, Wagner JD, Wenck S, Johnson CS, Coleman JJ 3rd. The prognostic importance of sentinel lymph node biopsy in thin melanoma. Ann Surg Oncol. 2006 Jul;13(7):927-32. doi: 10.1245/ASO.2006.04.023. Epub 2006 May 22. PMID 16788753
- [Background] Sandru A, Voinea S, Panaitescu E, Blidaru A. Survival rates of patients with metastatic malignant melanoma. J Med Life. 2014 Oct-Dec;7(4):572-6. PMID 25713625
- [Background] Tsao H, Atkins MB, Sober AJ. Management of cutaneous melanoma. N Engl J Med. 2004 Sep 2;351(10):998-1012. doi: 10.1056/NEJMra041245. No abstract available. PMID 15342808
- [Background] Hersey P, Gallagher S. Intralesional immunotherapy for melanoma. J Surg Oncol. 2014 Mar;109(4):320-6. doi: 10.1002/jso.23494. Epub 2013 Dec 3. PMID 24301265
- [Background] Sloot S, Rashid OM, Sarnaik AA, Zager JS. Developments in Intralesional Therapy for Metastatic Melanoma. Cancer Control. 2016 Jan;23(1):12-20. doi: 10.1177/107327481602300104. PMID 27009452
- [Background] Boyd KU, Wehrli BM, Temple CL. Intra-lesional interleukin-2 for the treatment of in-transit melanoma. J Surg Oncol. 2011 Dec;104(7):711-7. doi: 10.1002/jso.21968. Epub 2011 Jul 8. PMID 21744347
- See also: New treatments for metastatic melanoma — http://www.skincancer.org/skin-cancer-information/melanoma/melanoma-treatments/treatment-of-metastatic-melanoma

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intralesional IL-2 Injection | Saline Injection
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Total baseline participants n=1
Groups:
- Total: Total of all reporting groups
Arm/Group | Intralesional IL-2 Injection | Saline Injection | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Number of Patients Needed to Obtain Significance
Description: Data will be analyzed in order to achieve a statistically significant differentiation between treatment and control outcomes in study measures including tumor infiltrating lymphocytes (TILs) and circulating immunomodulators.
Time Frame: 1 year
Population: Data were not collected for tumor infiltrating lymphocytes (TILs) and circulating immunomodulators because patient was lost to follow-up.
Arm/Group | Intralesional IL-2 Injection | Saline Injection
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Assessment of Metastasis
Description: All patients will receive assessments every 4 months for 2 years and then biannual assessments for years 3-5 after the initial intervention to assess disease metastasis in treatment and control groups. Both number of new metastases (integer value) and thickness (mm) will be measured as a part of this assessment.
Time Frame: Assessments every 4 months for 2 years. Biannual assessments for years 3-5.
Population: Assessment of new metastases data could not be collected as patient was lost to follow-up.
Arm/Group | Intralesional IL-2 Injection | Saline Injection
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Assessment of RNA Genetic Profile
Description: RNA analysis of excised tissue will be compared to unaffected patient tissue obtained from the clear margins of the excisional biopsy to assess genetic changes resulting from the melanoma and treatment/placebo injections.
Time Frame: RNA analysis of excised tissue up to 5 years.
Population: Data were not collected for RNA analysis because patient was lost to follow-up.
Arm/Group | Intralesional IL-2 Injection | Saline Injection
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Assessment of Systemic Immune Response: Proteomic Analysis
Description: Proteomic analysis will be conducted on blood samples to assess systemic immune response to both treatment and control groups. Serum collected from patient blood samples will be used for proteomic analysis to assess protein expression, including circulating immunomodulators (cytokines and chemokines) before, and after, treatment. This study may serve to help develop diagnostic protocols and methods of assessing response to treatments.
Time Frame: Proteomic analysis of serum samples up to 5 years
Population: Data were not collected for proteomic analysis because patient was lost to follow-up.
Arm/Group | Intralesional IL-2 Injection | Saline Injection
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Assessment of Systemic Immune Response: Metabolomic Analysis
Description: Metabolomic analysis will be conducted on urine samples to assess systemic immune response to both treatment and control groups. All tumor and tissue produce by products in waste that are excreted by the kidneys. Urine samples can be evaluated using techniques, such as Mass Spectrometric, to determine if biological compounds can be identified in association with the presence of a malignant process that would not be produced by normal tissue.This study may serve to help develop diagnostic protocols and methods of assessing response to treatments.
Time Frame: Metabolomic analysis of urine samples up to 5 years
Population: Data were not collected for metabolomic analysis because patient was lost to follow-up.
Arm/Group | Intralesional IL-2 Injection | Saline Injection
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: 1
Arm/Group | Intralesional IL-2 Injection | Saline Injection
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/28/NCT03233828/Prot_SAP_004.pdf